CLINICAL TRIAL: NCT04543708
Title: Treatment of Tonsillar Abscess: A Randomized Clinical Trial in a Tertiary Center
Brief Title: Surgical Treatment of Tonsillar Abscess
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, François Voruz, Principal investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01516
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Tonsillar Abscess
Keywords: Tonsil; Abscess; Tonsillectomy; Local anesthesia; CT-scan
MeSH Terms: conditions — Abscess | interventions — Tonsillectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incision drainage (Active Comparator): Adult with clinical suspicion of tonsillar abscess who underwent a CT-scan confirming the abscess will be randomly assigned to one arm or the other. "Incision drainage" arm will benefit from drainage of the tonsillar abscess under local anesthesia and then be hospitalized for intravenous antibiotics. If the incision drainage fails, they will get a tonsillectomy under general anesthesia.
  Interventions: Procedure: Incision drainage
- Tonsillectomy (Active Comparator): Adult with clinical suspicion of tonsillar abscess who underwent a CT-scan confirming the abscess will be randomly assigned to one arm or the other. "Tonsillectomy" arm will benefit from tonsillectomy under general anesthesia and then be hospitalized for intravenous antibiotics.
  Interventions: Procedure: Tonsillectomy

INTERVENTIONS:
Procedure: Incision drainage — Oropharyngeal pre-anesthesia is performed with 10% xylocaine spray, then submucosal anesthesia of the anterior pillar of the tonsil is performed with 2 ml of Rapidocaine or Rapidocaine 1 or 2% adrenaline. A scalpel incision is made with the search for the abscess pocket with a crile. If pus is present, a NaCl / Betadine rinse is performed. A syringe puncture can help locate the abscess if needed. The duration is approximately 15 minutes.
  If no purulent pouch is found, the procedure is completed with tonsillectomy under general anesthesia.
  Arms: Incision drainage
Procedure: Tonsillectomy — Under general anesthesia, in dorsal decubitus, an autostatic mouth opener is placed, an incision of the anterior pillar of the tonsil allows the opening of the capsular space, along which the entire tonsil is dissected until complete extraction, hemostasis is performed, then the patient is awakened. The duration is approximately 30 minutes.
  Arms: Tonsillectomy

SUMMARY:
The diagnosis and treatment of tonsillar abscess are very physician-dependent, as sufficient prospective medical literature is lacking to choose the most efficient regimen. The proposed study aims to assess the therapeutic efficacy of tonsillectomy compared to drainage under local anesthesia. This is a prospective, randomized clinical trial in adults in a tertiary care center in Geneva (Switzerland).

DETAILED DESCRIPTION:
Introduction:

Tonsillar abscess is the most common complication of acute bacterial angina. The abscess is located in the majority of cases in the capsular space and occasionally within the tonsil itself. The ethiopathogenesis is polymicrobial, composed mainly of Streptococcus Pyogenes (aerobic) and Fusobacterium Necrophorum (anaerobe). This condition mainly affects young adults, smokers and significantly impacts quality of life. Symptoms are noisy, characterized by severe odynodysphagia, often limited mouth opening (trismus), and occasionally dyspnea, fever, and decreased general condition. Its complications include upper airway obstruction, spread of infection into the deep tissues of the neck and mediastinum, septic venous thrombosis, and arterial hemorrhage from contact necrosis. The descriptions of the management of this pathology are centuries old, but even today there is a need to drain the pus. We estimate that around 200 patients per year present to our University Hospital in Geneva (Switzerland) with suspected tonsillar abscess.

Diagnosis:

The medical literature describes several diagnostic methods without clear consensus on the most effective. The doctor's clinical suspicion varies according to the examiner's experience, although certain criteria are recognized as good predictors of the presence of an abscess (trismus, edema, uvula deviation, "hot potato voice", reflex otalgia), but with limited sensitivity and specificity. When clinically suspected, confirmation of the presence of pus can be determined by direct puncture or drainage, allowing immediate diagnosis, but with a high proportion of false negatives and requiring a painful invasive procedure. Ultrasound (US) and Computed Tomography (CT) provide a painless diagnosis, but US requires a specific oral probe and may be unfeasible in case of trismus, and its interpretation is very examiner-dependent. CT remains an irradiating, costly and time-consuming exam, but it is sensitive and can formally exclude any associated complication (venous thrombosis, retro- or parapharyngeal extension, contralateral involvement). The gold-standard for the diagnosis of a tonsillar abscess is the direct visualization of pus during drainage.

Treatment:

Regarding the treatment, here too the evidence-based literature is not clear about the most effective (except in children, in whom local anesthesia intervention is most of the time impractical). It usually consists of a combination of medical and surgical therapy. Medical therapy generally includes - in addition to hydration and pain-killers - intravenous antibiotics and requires approximately 3 days of hospitalization. There are several described technics for the surgical drainage. Repeated needle punctures, incisional drainage under local anesthesia, and tonsillectomy under general anesthesia. The latter two are favored because they are more effective on immediate pain. To our knowledge, only two prospective randomized studies (partially for one) of 51 and 53 patients have studied the efficacy of these two interventions and their conclusions only relate to the absence of difference in the length of hospital stay.

The retrospective data show good efficacy of both modalities (incision drainage under local anesthesia vs tonsillectomy under general anesthesia) and the choice of their execution is strongly center- and physician-dependent. Incision drainage avoids general anesthesia but is extremely unpleasant, requiring repeated rinsing which is painful for the patient and time-consuming for the medical team. This modality is grafted with a failure rate of around 20% in the literature as well as in our own experience, requiring further tonsillectomy under general anesthesia. Furthermore, the recurrence rate is estimated at 9-22%. Conversely, the first-line tonsillectomy requires a general anesthesia but immediately relieves some of the pain and the trismus, allows an almost certain resolution of the infection, prevents any recurrence, seems economically more advantageous and does not require the collaboration of the patient during the procedure.

As the medical literature does not offer clear guidelines based on prospective trials, the proposed study aims to prospectively evaluate the therapeutic efficacy of the tonsillectomy compared to the drainage under local anesthesia.

This is a prospective, randomized clinical trial by adults in a tertiary care center in Geneva (Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age with clinical suspicion of unilateral tonsillar abscess without signs of "extra-capsular" complication.
* Obtaining informed consent.

Exclusion Criteria:

* Contraindications to injected CT or drainage in local anesthesia (allergy to iodinated contrast product, allergy to local anesthetics, phobia of needles, major trismus).
* Parapharyngeal or retropharyngeal abscess, or associated venous thrombosis found on CT.
* Imminent threat to the upper respiratory tract (glottic edema, acute dyspnea).
* Inability to understand the different procedures (dementia, impossible communication, substance abuse).
* Anamnestic pregnancy.
* Antiaggregant or anticoagulant treatment.
* Treatment of corticosteroids during the management of emergencies and in hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of treatment success (%) | 3 days
  Disappearance of fever if any + decrease in leukocytosis and CRP value + no sign of recollection nor cervical extension of the infection.

SECONDARY OUTCOMES:
Recurrence rate (%) | 3 and 12 months
  Reccurence of a tonsillar abscess on the same side post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: François Voruz, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospitalas Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Powell EL, Powell J, Samuel JR, Wilson JA. A review of the pathogenesis of adult peritonsillar abscess: time for a re-evaluation. J Antimicrob Chemother. 2013 Sep;68(9):1941-50. doi: 10.1093/jac/dkt128. Epub 2013 Apr 23. PMID 23612569
- [Background] Windfuhr JP, Toepfner N, Steffen G, Waldfahrer F, Berner R. Clinical practice guideline: tonsillitis II. Surgical management. Eur Arch Otorhinolaryngol. 2016 Apr;273(4):989-1009. doi: 10.1007/s00405-016-3904-x. Epub 2016 Feb 16. PMID 26882912
- [Background] Albertz N, Nazar G. Peritonsillar abscess: treatment with immediate tonsillectomy - 10 years of experience. Acta Otolaryngol. 2012 Oct;132(10):1102-7. doi: 10.3109/00016489.2012.684399. Epub 2012 Jun 18. PMID 22708633
- [Background] Lehnerdt G, Senska K, Fischer M, Jahnke K. [Smoking promotes the formation of peritonsillar abscesses]. Laryngorhinootologie. 2005 Sep;84(9):676-9. doi: 10.1055/s-2005-870289. German. PMID 16142623
- [Background] Powell J, Powell EL, Conroy K, Hopkins C, Moor JW, Wilson JA. Throat-related quality of life in peritonsillar abscess sufferers: application of the adult tonsil outcome inventory. J Laryngol Otol. 2013 Dec;127(12):1190-3. doi: 10.1017/S0022215113003071. Epub 2013 Nov 20. PMID 24252628
- [Background] Grant MC, Raggio B, Barton B, Guarisco JL. Establishing the Need for an Evidence-Based Treatment Algorithm for Peritonsillar Abscess in Children. Clin Pediatr (Phila). 2018 Oct;57(12):1385-1390. doi: 10.1177/0009922818778048. Epub 2018 May 29. PMID 29808740
- [Background] Scott PM, Loftus WK, Kew J, Ahuja A, Yue V, van Hasselt CA. Diagnosis of peritonsillar infections: a prospective study of ultrasound, computerized tomography and clinical diagnosis. J Laryngol Otol. 1999 Mar;113(3):229-32. doi: 10.1017/s0022215100143634. PMID 10435129
- [Background] Salihoglu M, Eroglu M, Yildirim AO, Cakmak A, Hardal U, Kara K. Transoral ultrasonography in the diagnosis and treatment of peritonsillar abscess. Clin Imaging. 2013 May-Jun;37(3):465-7. doi: 10.1016/j.clinimag.2012.09.023. Epub 2012 Oct 25. PMID 23102927
- [Background] Carratola MC, Frisenda G, Gastanaduy M, Guarisco JL. Association of Computed Tomography With Treatment and Timing of Care in Adult Patients With Peritonsillar Abscess. Ochsner J. 2019 Winter;19(4):309-313. doi: 10.31486/toj.18.0168. PMID 31903053
- [Background] Patel KS, Ahmad S, O'Leary G, Michel M. The role of computed tomography in the management of peritonsillar abscess. Otolaryngol Head Neck Surg. 1992 Dec;107(6 Pt 1):727-32. doi: 10.1177/019459988910700603.1. PMID 1470448
- [Background] Teschner M, Aljeraisi T, Giesemann A, Gotz F, Lenarz T, Kontorinis G. [The role of CT in the diagnosis of peritonsillar abscesses after Punctio Sicca]. Laryngorhinootologie. 2013 Jan;92(1):25-9. doi: 10.1055/s-0032-1327709. Epub 2012 Nov 19. German. PMID 23165703
- [Background] Johnson RF, Stewart MG, Wright CC. An evidence-based review of the treatment of peritonsillar abscess. Otolaryngol Head Neck Surg. 2003 Mar;128(3):332-43. doi: 10.1067/mhn.2003.93. PMID 12646835
- [Background] Powell J, Wilson JA. An evidence-based review of peritonsillar abscess. Clin Otolaryngol. 2012 Apr;37(2):136-45. doi: 10.1111/j.1749-4486.2012.02452.x. PMID 22321140
- [Background] Hur K, Zhou S, Kysh L. Adjunct steroids in the treatment of peritonsillar abscess: A systematic review. Laryngoscope. 2018 Jan;128(1):72-77. doi: 10.1002/lary.26672. Epub 2017 May 31. PMID 28561258
- [Background] Fagan JJ, Wormald PJ. Quinsy tonsillectomy or interval tonsillectomy--a prospective randomised trial. S Afr Med J. 1994 Oct;84(10):689-90. PMID 7839259
- [Background] Chowdhury CR, Bricknell MC. The management of quinsy--a prospective study. J Laryngol Otol. 1992 Nov;106(11):986-8. doi: 10.1017/s002221510012153x. PMID 1479277
- [Background] Yung AK, Cantrell RW. Quinsy tonsillectomy. Laryngoscope. 1976 Nov;86(11):1714-7. doi: 10.1288/00005537-197611000-00015. PMID 1068337
- [Background] Clerc S, Soldati D. [Socioeconomic aspects in the therapy of peritonsillar absscess]. Schweiz Med Wochenschr. 2000;Suppl 125:17S-19S. French. PMID 11141930
- [Derived] Voruz F, Revol R, Mermod M, Senn P, Monnier Y, Dulguerov N. A randomized clinical trial of peritonsillar abscess treatment comparing drainage and tonsillectomy. Am J Otolaryngol. 2025 Nov-Dec;46(6):104745. doi: 10.1016/j.amjoto.2025.104745. Epub 2025 Oct 20. PMID 41192203